CLINICAL TRIAL: NCT03495622
Title: Effectiveness of a Combined CHW and Text Messaging-based Tobacco Intervention in India Project MUKTI: A Multi-Unit Kit for Tobacco Intervention
Brief Title: Effectiveness of a Combined CHW and Text Messaging-based Tobacco Intervention in India
Acronym: MUKTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Richard Josephson, MS MD, Professor of Medicine Case Western Reserve University School of Medicine/ Director Cardiovascular and Pulmonary Rehabilitation program University Hospitals Cleveland Medical Center, Division of Cardiovascular Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-17-29
Record Dates: First submitted 2018-03-26; First posted 2018-04-12 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Smoking Cessation
Keywords: Text messaging; Community health worker; Smoking cessation; India; Cardiovascular mortality
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing/Text messaging (Experimental): Home visits by community health worker to deliver motivational interviewing and set up a structured text messaging strategy designed around a pre-determined quit date for smoking cessation.
  Interventions: Behavioral: Motivational Interviewing/Text messaging
- Control (No Intervention): All participants will receive brief verbal advice about the hazards of smoking and the benefits of smoking cessation.

INTERVENTIONS:
Behavioral: Motivational Interviewing/Text messaging — The intervention is a multi-component one that is tailored to the individual and will target smoking cessation. The CHW, after identifying the individual's stage of behavior change, will provide motivational interviewing and set up an automatic text messaging system with their mobile phones that are structured around a quit date chosen by the participant.
  The CHW visits are pre-determined and she monitors the progress of the individual regularly. She may restart the process of determining the stage of behavior change for those who relapse or quit the intervention midway thereby reassigning them to the appropriate phase of the trial
  Arms: Motivational Interviewing/Text messaging

SUMMARY:
The study is a multi-center 1-year community-based cluster randomized controlled trial to assess the role of a combined community health worker and mobile health intervention in controlling one of the most common cardiovascular risk factors, tobacco use. Participants will include 560 adults, 18-70 years of age, from the urban communities of Dalkhola, West Bengal, and Jabalpur, Madhya Pradesh, India. The hypothesis of the study is that this combined approach can result in increased quit rate among tobacco users.

DETAILED DESCRIPTION:
Smoking tobacco is a major contributor to the global cardiovascular disease burden. India bears a huge part of this burden and it is estimated that nearly a quarter million individuals aged >15 years consume tobacco in India. Moreover, about 70% of tobacco deaths are reported to be in the age range of 30-69 years.

Motivational interviewing (MI) is an innovative manner of communication which puts the focus on the patient and strengthens their motivation for behavior change without overt confrontation or persuasion. MI delivered by community health workers (CHW) is part of the strategy planned by the investigators.

In order to deliver personalized assistance and increase penetration of the required intervention into different parts of the country, text messaging is a promising strategy in low and middle-income countries but there is no data regarding its application for tobacco use in India.

The investigators plan to screen 560 individuals between the age of 18 and 70 years for smoking from 16 randomly selected clusters in the economically backward urban towns of Dalkhola (West Bengal) and Jabalpur (Madhya Pradesh). The screening will be done using house to house visits by CHWs who will administer a questionnaire based on the WHO STEPS survey. An individual identified as a chronic tobacco user irrespective of his/her stage of behavior change will be eligible for further participation in the study and assigned to the appropriate intervention arm. Clusters will be randomized to either receive the combined intervention or usual care.

Apart from screening and recruitment, CHWs will be responsible for differentiating individuals between being pre-contemplative vs contemplative. Based on their readiness to quit, participants will receive a structured intervention which involves motivational interviewing delivered by the CHW in their homes and weekly support provided through regular mobile text messages.

The CHWs will be chosen from the study population based on a set of criteria through a formal selection panel after consulting with the local leaders and physicians. They will undergo a week of training for the screening process, an additional week for the intervention and finally a refresher course every 6 months.

The text messages are selected from a pre-determined database of messages and the content of which changes based on the individual's stage of behavior change. The messages are delivered automatically every other day of the week and are controlled by the investigators in Cleveland, Ohio, USA.

The control group, during their screening visit, will be informed of their problems, given a brief pamphlet and encouraged to seek physician help.

The investigators hypothesize that a community health worker based intervention, utilizing motivational interviewing and health education, coupled with text messaging based support will lead to increased quit rates amongst participants who are daily smokers.

At the end of one year, the self-reported abstinence of the participants in the intervention arm will be recorded and biochemically verified with a carbon monoxide breath analyzer test.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 18 and 70 years, who smoke cigarettes or bidis daily
2. Individuals able and willing to give informed consent

Exclusion Criteria:

1. Individuals who are bed-bound because of acute illness or have a chronic condition that makes them bed-bound.
2. Individuals who refuse consent
3. Individuals who do not reside in the community and are only visiting, therefore being unlikely to be available for continuous follow up. Individuals who have stayed less than 6 months in the study area, or whose name is not on the voter list of the area will be excluded.
4. Individuals who are not able to participate in the intervention due to significant disabilities, such as blindness, deafness or the intellectually disabled. This determination is at the discretion of the community health worker.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Quit rate at the end of 1 year | 1 year
  Self-reported abstinence, biochemically verified, for the past 14 days at the end of 1 year from the start of the intervention.

SECONDARY OUTCOMES:
Relapse rate at the end of 1 year | 1 year
  The number of individuals who have relapsed into smoking after completing the intervention at the end of 1 year.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - SEHAT, Jabalpur, Madhya Pradesh
  - SEHAT, Dalkhola, West Bengal

IPD SHARING:
Plan to Share IPD: Undecided